CLINICAL TRIAL: NCT05732883
Title: The Use of Dexamethasone in Total Thyroidectomy to Improve Voice Outcome and Hypocalcaemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tseung Kwan O Hospital, Hong Kong (Other)
Collaborators: United Christian Hospital (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, YEUNG WING CHI ZENON, Associate Consultant, Department of Otorhinolaryngology, Head and Neck Surgery, Tseung Kwan O Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KC/KE-22-0022/FR-4
Record Dates: First submitted 2022-12-27; First posted 2023-02-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Voice Change; Hypocalcemia
Keywords: Voice dysfunction; Hoarseness of Voice; Vocal cord palsy; Hypocalcemia; Hypoparathyroidism; Thyroidectomy; Dexamethasone; Steroid
MeSH Terms: conditions — Dysphonia; Hypocalcemia; Hoarseness; Vocal Cord Paralysis; Hypoparathyroidism | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multi-specialty, double-blind, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, randomized, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone group (Experimental): One dose of 8mg in 2ml Dexamethasone will be given
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): One dose of 2ml 0.9% Normal saline will be given
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone injection
  Arms: Dexamethasone group
Drug: Normal saline — Placebo
  Arms: Placebo group

SUMMARY:
Thyroidectomy is a standard procedure for benign and malignant pathologies of the thyroid gland. Each year, some 100 total thyroidectomies are performed in Kowloon East Cluster, Hospital Authority, Hong Kong. Total thyroidectomy is associated with voice dysfunction and temporary hypocalcaemia in up to 80% and 50%, respectively. Previous study from our institute showed a 3% rate of permanent vocal cord palsy and 16% of permanent hypoparathyroidism requiring calcium and/or vitamin D supplements. The use of dexamethasone has been studied in the past in total thyroidectomy patients and has been shown to be safe and effective in improving post-operative nausea and vomiting. No complications or drug related side effects were associated with a single dose of steroid. Recent studies have also shown that Dexamethasone is effective in improving voice outcome and hypocalcaemia in thyroidectomy patients. The investigators aim to study the effect of Dexamethasone in post-operative voice outcome and hypocalcaemia. Objective assessment of the vocal cords during phonation will be performed pre-operative and post-operatively. Serum Calcium level will be monitored.

DETAILED DESCRIPTION:
This is a multi-specialty, double-blind, randomized, placebo-controlled trial involving the Departments of Surgery in United Christian Hospital, Tseung Kwan O Hospital and Department of Ear, Nose and Throat, United Christian Hospital and Tseung Kwan O Hospital, Kowloon East Cluster. The primary objective is to investigate the effect of Dexamethasone in post-operative voice outcome and hypocalcaemia in total thyroidectomy patients. The secondary outcome aims to investigate the mechanism of voice dysfunction in thyroidectomy patients using objective assessment tools.

To streamline the practice among various departments and to minimize any potential confounders, the peri-operative anaesthetic and post-operative analgesic protocols are standardized. The surgical techniques are also standardized using capsular dissection with positive identification and preservation of the recurrent laryngeal nerve.

Patient's voice and vocal cord mobility will be assessed pre-operatively and post-operatively. Objective assessment of the vocal cord will be carried out using video stroboscopy to document the mobility, waveform and vibration, symmetry and any arytenoid abnormality. Subjective and objective assessment of the voice outcome will be conducted by speech therapists using standardized voice assessment protocol. The trend of hypocalcaemia (Calcium level and parathyroid hormone level) will be monitored and correlated with the use of Dexamethasone. Possible side effect (e.g. wound infection) from the use of Dexamethasone will be analysed

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Patients undergoing total thyroidectomy for benign pathologies
* MNG
* Toxic nodular goitre
* Graves' disease

Exclusion Criteria:

* Non-communicable patients
* Patients contraindicated for steroid (DM, Hepatitis carrier, Tuberculosis, peptic ulcer disease)
* Patients contraindicated for analgesics including Panadol, Celebrex, Tramadol or Levobupivacaine
* Malignant thyroid disease
* Patients with previous thyroid surgery, or neck surgery
* Pre-existing hoarseness of voice of any cause or pre-existing vocal cord palsy
* Pregnancy / Lactating female patients
* Pre-existing renal disease / autoimmune disease on steroids
* Patients who require steroid cover during operation e.g. hydrocortisone perioperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative calcium and parathyroid hormone level on POD1 | Post-op 1 day
  Serum calcium and parathyroid hormone level will be monitored
Post-operative calcium and parathyroid hormone level after 3 months post-op | Post-op 3 months
  Serum calcium and parathyroid hormone level will be monitored
Post-operative calcium and parathyroid hormone level after 6 months post-op | Post-op 6 months
  Serum calcium and parathyroid hormone level will be monitored
Voice Handicap Index (VHI-10) | Post-op 1 week
  Subjective voice assessment consisting of 10 questions. Each question 0-4 score
Voice Handicap Index (VHI-10) | Post-op 3 months
  Subjective voice assessment consisting of 10 questions. Each question 0-4 score
Voice Handicap Index (VHI-10) | Post-op 6 months
  Subjective voice assessment consisting of 10 questions. Each question 0-4 score
Perceptual Evaluation: Cantonese Perceptual Evaluation of Voice (CanPEV) | Post-op 1 week
  Objective voice assessment consisting of 10 questions. Each question 1-10 score. 1 being normal and 10 being the most severe voice dysfunction
Perceptual Evaluation: Cantonese Perceptual Evaluation of Voice (CanPEV) | Post-op 3 months
  Objective voice assessment consisting of 10 questions. Each question 1-10 score. 1 being normal and 10 being the most severe voice dysfunction
Perceptual Evaluation: Cantonese Perceptual Evaluation of Voice (CanPEV) | Post-op 6 months
  Objective voice assessment consisting of 10 questions. Each question 1-10 score. 1 being normal and 10 being the most severe voice dysfunction
Acoustic Evaluation | Post-op 1 week
  Instruct patient to sustain vowel /a/ and to read aloud the Hong Kong passage at a comfortable pitch and loudness level for about 3-5 seconds. Keep a distance of 15cm from the microphone for recording. Highlight the middle 3 seconds for analysis. To assess the fundamental frequency (Hz) and performance (dB)
Acoustic Evaluation | Post-op 3 months
  Instruct patient to sustain vowel /a/ and to read aloud the Hong Kong passage at a comfortable pitch and loudness level for about 3-5 seconds. Keep a distance of 15cm from the microphone for recording. Highlight the middle 3 seconds for analysis. To assess the fundamental frequency (Hz) and performance (dB)
Acoustic Evaluation | Post-op 6 months
  Instruct patient to sustain vowel /a/ and to read aloud the Hong Kong passage at a comfortable pitch and loudness level for about 3-5 seconds. Keep a distance of 15cm from the microphone for recording. Highlight the middle 3 seconds for analysis. To assess the fundamental frequency (Hz) and performance (dB)
Aerodynamic Evaluation (Maximum sustained phonation) | Post-op 1 week
  Instruct patient to sustain vowel /a/ at a comfortable pitch and loudness level for as long as possible after taking a deep breath. Recorded in seconds
Aerodynamic Evaluation (Maximum sustained phonation) | Post-op 3 months
  Instruct patient to sustain vowel /a/ at a comfortable pitch and loudness level for as long as possible after taking a deep breath. Recorded in seconds
Aerodynamic Evaluation (Maximum sustained phonation) | Post-op 6 months
  Instruct patient to sustain vowel /a/ at a comfortable pitch and loudness level for as long as possible after taking a deep breath. Recorded in seconds

SECONDARY OUTCOMES:
Calcium and Rocaltrol requirement | Post-op 1 week
  The required dosage of Calcium Carbonate and Rocaltrol will be documented
Calcium and Rocaltrol requirement | Post-op 3 months
  The required dosage of Calcium Carbonate and Rocaltrol will be documented
Calcium and Rocaltrol requirement | Post-op 6 months
  The required dosage of Calcium Carbonate and Rocaltrol will be documented
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Post-op 1 week
  Number of participants experiencing side effects from Dexamethasone will be documented
Stroboscopic Assessment (Vocal Fold Edge) | Post-op 1 week
  Score 1-5 (1 - Smooth and straight; 5 - Rough and irregular)
Stroboscopic Assessment (Vocal Fold Edge) | Post-op 3 months
  Score 1-5 (1 - Smooth and straight; 5 - Rough and irregular)
Stroboscopic Assessment (Vocal Fold Edge) | Post-op 6 months
  Score 1-5 (1 - Smooth and straight; 5 - Rough and irregular)
Stroboscopic Assessment (Glottic Closure) | Post-op 1 week
  Grading 1-7 (1. Complete 2. Anterior chink 3. Irregular 4. Bowing 5.Posterior chink 6. Hourglass 7 Incomplete)
Stroboscopic Assessment (Glottic Closure) | Post-op 3 months
  Grading 1-7 (1. Complete 2. Anterior chink 3. Irregular 4. Bowing 5.Posterior chink 6. Hourglass 7 Incomplete)
Stroboscopic Assessment (Glottic Closure) | Post-op 6 months
  Grading 1-7 (1. Complete 2. Anterior chink 3. Irregular 4. Bowing 5.Posterior chink 6. Hourglass 7 Incomplete)
Stroboscopic Assessment (Vertical Level of Approximation) | Post-op 1 week
  1 - Equal 2 - Right lower 3 - Left lower 4 - Questionable
Stroboscopic Assessment (Vertical Level of Approximation) | Post-op 3 months
  1 - Equal 2 - Right lower 3 - Left lower 4 - Questionable
Stroboscopic Assessment (Vertical Level of Approximation) | Post-op 6 months
  1 - Equal 2 - Right lower 3 - Left lower 4 - Questionable
Stroboscopic Assessment (Amplitude) | Post-op 1 week
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - No visible movement
Stroboscopic Assessment (Amplitude) | Post-op 3 months
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - No visible movement
Stroboscopic Assessment (Amplitude) | Post-op 6 months
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - No visible movement
Stroboscopic Assessment (Mucosal wave) | Post-op 1 week
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - Absent
Stroboscopic Assessment (Mucosal wave) | Post-op 3 months
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - Absent
Stroboscopic Assessment (Mucosal wave) | Post-op 6 months
  1 - Normal 2 - Slightly decreased 3 - Moderately decreased 4 - Severely decreased 5 - Absent
Stroboscopic Assessment (Regularity) | Post-op 1 week
  1 - Regular 2 - Sometimes irregular 3 - Most irregular 4 - Always irregular
Stroboscopic Assessment (Regularity) | Post-op 3 months
  1 - Regular 2 - Sometimes irregular 3 - Most irregular 4 - Always irregular
Stroboscopic Assessment (Regularity) | Post-op 6 months
  1 - Regular 2 - Sometimes irregular 3 - Most irregular 4 - Always irregular
Stroboscopic Assessment (Ventricular folds) | Post-op 1 week
  Movement - 1.Normal 2.Slight compress 3.Moderate compress 4.Full compress
Stroboscopic Assessment (Ventricular folds) | Post-op 3 months
  Movement - 1.Normal 2.Slight compress 3.Moderate compress 4.Full compress
Stroboscopic Assessment (Ventricular folds) | Post-op 6 months
  Movement - 1.Normal 2.Slight compress 3.Moderate compress 4.Full compress

CONTACTS AND LOCATIONS:
Overall Officials: Jason YK Chan, MBBS, Study Director — Department of Otorhinolaryngology, Head and Neck Surgery, The Chinese University of Hong Kong; Zenon YEUNG, MbChB, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery, The Chinese University of Hong Kong
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, United Christian Hospital and Tseung Kwan O Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No